CLINICAL TRIAL: NCT01066585
Title: A Double-Blind Randomized Study to Compare the Efficacy, Safety and Local Tolerability of a 0.5% Ivermectin Cream Compared to a Topical Vehicle Control in Subjects With Pediculus Humanus Capitis Infestation
Brief Title: A Safety and Efficacy Study Comparing 0.5% Ivermectin Cream to a Vehicle Control in Subjects With Head Lice Infestation
Acronym: LICE OUT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Topaz Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOP011
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Results first posted 2012-04-04 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Head Lice
Keywords: Head lice; Pediculus humanus capitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.5% Ivermectin Cream (Experimental)
  Interventions: Drug: Ivermectin Cream
- Vehicle control (Placebo Comparator)
  Interventions: Drug: vehicle control

INTERVENTIONS:
Drug: Ivermectin Cream — Up to 4 ounces of topical 0.5% Ivermectin Cream applied to the hair and scalp on day 1
  Arms: 0.5% Ivermectin Cream
Drug: vehicle control — Up to 4 ounces of vehicle control applied to the hair and scalp on day 1
  Arms: Vehicle control

SUMMARY:
The purpose of this study is to determine if 0.5% Ivermectin Cream is a safe and effective treatment for head lice infestations.

ELIGIBILITY:
Inclusion Criteria:

* Index subjects must have an active head lice infestation defined as: At least 3 live lice (adults and/or nymphs) present on the scalp and/or hair, as determined by a trained evaluator. The index subject must be the youngest family member presenting with at least 3 live lice. After the index subject has been identified, additional infested household members (see b below) will be enrolled.
* Household subjects must have an active head lice infestation defined as: At least 1 live louse (adult and/or nymph) present on the scalp and/or hair, as determined by a trained evaluator (with the exception of the male head of household who may self-assess as being lice free).
* Subject is male or female.
* Subject is at least 6 months of age at time of enrollment.
* Subject is in good general health based on medical history.
* Each subject must have an appropriately signed Informed Consent agreement. A caregiver must sign an Informed Consent agreement for children not old enough to do so. Children of a specified age will be administered a child's assent form.
* The caregiver of a subject must be willing to allow all household members to be screened for head lice. If other household members are found to have an active head lice infestation, according to the criteria b (above), they must be willing and able to participate in the study. No more than one working male per household may be excluded from evaluation if he is assessed as being lice free by himself or the caregiver and cannot come in due to his work schedule. If this individual may have lice, he must come to the test facility; otherwise the entire household will be excluded from study participation.
* Subject and/or their caregiver must be physically able and willing to apply the test article.
* Subject agrees not to use any other form of lice treatments (commercial, community-anecdotal, or mechanical/manual) while participating in the study.
* Following application and rinsing of the test article, subject agrees not to shampoo, wash, or rinse their hair or scalp until the 24-hour post-treatment evaluation has been completed.
* Subject agrees to not cut or chemically treat their hair while participating in the study.
* Subject agrees to follow all study instructions.
* Female subjects of childbearing potential (including a female caregiver even if she is not being treated) must be willing to have a urine pregnancy test.
* In the event of a subject judged to be incapable of self-treating, the household must have a caregiver willing to apply the treatment at home.

Exclusion Criteria:

* History of irritation or sensitivity to ivermectin or the cream components, pediculicides or hair care products.
* Presentation at the treatment site with visible skin/scalp condition(s) that are not attributable to head lice infestation, such as an erythema score that is >2, blisters, vesicles which, in the opinion of the investigative personnel or sponsor, will interfere with safety and/or efficacy evaluations.
* Presentation at the treatment site with eczema or atopic dermatitis.
* Treatment for head lice (Over the counter [OTC], home remedy and/or Prescription) in the last 7 days.
* Any condition or illness that, in the opinion of the investigator, may compromise the objective of the protocol.
* Is receiving any other treatment which, in the opinion of the investigator or study monitor, may interfere with the study results.
* Females (including caregivers who come in contact with the investigational product) who are pregnant, nursing or planning a pregnancy. (NOTE: female caregivers and all enrolled females of childbearing potential must have a negative urine pregnancy test prior to treatment). If a household has a pregnant female who has an active case of lice, the entire household is excluded from participation. If this pregnant household member does not have an active infestation, this individual must NOT be the caregiver (one who provides treatment to other household members).
* Is of child-bearing potential and unwilling to use an adequate method of contraception for the duration of the study. Adequate methods of contraception include: abstinence, vasectomized partner, oral birth control pills, birth control injections or patches, Intra uterine devices, condoms with a spermicidal jelly or a diaphragm with spermicidal jelly, surgical sterilization.
* Participation in a previous investigational drug study within the past 30 days.
* Prior participation in any ivermectin trials.
* Does not understand the requirements for study participation and/or may likely exhibit poor compliance, in the opinion of the investigator.
* Does not have a known household affiliation with their household members (i.e., do not stay in one household consistently, sleeping at one place several nights and then at another place or location). Household is defined as living in a shared area or space (for example the same house or apartment unit).

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Sanofi Topaz
Locations (8):
- United States (8):
  - Cactus Kids Pediatrics, Yuma, Arizona
  - Universal Biopharma Research, Inc, Dinuba, California
  - Lice Source Services, Inc., Plantation, Florida
  - LSRN, West Palm, Florida
  - Spence Medical Research, Picayune, Mississippi
  - Hill Top Research, Miamiville, Ohio
  - McKenzie Medical Center, McKenzie, Tennessee
  - Virginia Clinical Research, Inc., Norfolk, Virginia

REFERENCES:
- [Derived] Pariser DM, Meinking TL, Bell M, Ryan WG. Topical 0.5% ivermectin lotion for treatment of head lice. N Engl J Med. 2012 Nov 1;367(18):1687-93. doi: 10.1056/NEJMoa1200107. PMID 23113480

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and treated from 8 March 2010 to 9 June 2010 in 8 US clinical centers.
Pre-assignment Details: A total of 410 participants who met the inclusion and exclusion criteria were enrolled and treated.
Groups:
- 0.5% Ivermectin: Participants underwent a single treatment with 0.5% ivermectin cream at home on Day 1.
- Vehicle Control: Participants underwent a single treatment with vehicle control cream at home on Day 1.
Period: Overall Study
Arm/Group | 0.5% Ivermectin | Vehicle Control
Started | 211 | 199
Completed | 210 | 196
Not Completed | 1 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5% Ivermectin | Vehicle Control | Total
Number analyzed (Participants) | 211 | 199 | 410
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 164 | 149 | 313
  Between 18 and 65 years | 47 | 50 | 97
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 13.92 (12.00) | 15.05 (13.52) | 14.47 (12.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 164 | 336
  Male | 39 | 35 | 74
Region of Enrollment [Number; unit: Participants]
  United States | 211 | 199 | 410

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Index Participants Who Were Lice-Free by Day 2 That Were Maintained Through Day 15 Post-treatment With Either Ivermectin or Placebo (Vehicle Control)
Description: Treatment success defined as absence of live lice, was assessed in index participants, defined as the youngest person within each household who had at least 3 live lice present at Screening (Day 1). Treatment success was assessed by last observation carried forward (LOCF) imputation and treatment failure imputation.
Time Frame: Day 2 up to Day 15 post-application
Population: Treatment success was assessed in the Intent-to-treat population. Any participant with live lice on or after Day 2 received an FDA approved head lice treatment and was classified as a treatment failure, imputed as such for remaining assessments.
Measure: Number; unit: Percent of Participants
Arm/Group | 0.5% Ivermectin | Vehicle Control
Number analyzed (Participants) | 71 | 74
Percent of Participants
  Day 15 (LOCF Imputation) | 76 | 16 [0 to 0]
  Day 15 (Treatment Failure Imputation) | 76 | 15 [0 to 0]

2. Secondary Outcome: Percentage of All Participants Who Were Lice-Free by Day 2 That Were Maintained Through Day 15 Post-treatment With Either Ivermectin or Placebo (Vehicle Control)
Description: Treatment success, defined as absence of live lice, was assessed in all subjects. Treatment success was assessed by last observation carried forward (LOCF) imputation and treatment failure imputation.
Time Frame: Day 2 up to Day 15 post-application
Population: as for outcome 1
Measure: Number; unit: Percent of Participants
Arm/Group | 0.5% Ivermectin | Vehicle Control
Number analyzed (Participants) | 211 | 199
Percent of Participants
  Day 15 (LOCF Imputation) | 82 | 22 [0 to 0]
  Day 15 (Treatment Failure Imputation) | 81 | 21 [0 to 0]

3. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events Post-treatment With Either Ivermectin or Placebo (Vehicle Control)
Description: Severity of the adverse events were defined and classified as follows:
  'Mild' - Awareness of signs or symptoms, but easily tolerated; 'Moderate' - Discomfort to a degree that adverse event/adverse drug reaction causes interference with normal daily life activities and/or requires medication; 'Severe' - Incapacity with regard to work or usual daily life activities. Requires medical attention/intervention.
Time Frame: Day 1 up to Day 15 post-application.
Population: Adverse events were assessed in the Intent-to-treat (Safety) population.
Measure: Number; unit: Participants
Arm/Group | 0.5% Ivermectin | Vehicle Control
Number analyzed (Participants) | 210 | 199
Participants
  Any Lymphadenopathy | 0 | 1 [0 to 0]
  Severe Lymphadenopathy | 0 | 0 [0 to 0]
  Any Eye Irritation | 1 | 0 [0 to 0]
  Severe Eye Irritation | 0 | 0 [0 to 0]
  Any Impetigo | 0 | 1 [0 to 0]
  Severe Impetigo | 0 | 0 [0 to 0]
  Any Pharyngitis Streptococcal | 1 | 0 [0 to 0]
  Severe Pharyngitis Streptococcal | 0 | 0 [0 to 0]
  Any Tonsillitis | 1 | 0 [0 to 0]
  Severe Tonsillitis | 0 | 0 [0 to 0]
  Any Excoriation | 0 | 4 [0 to 0]
  Severe Excoriation | 0 | 0 [0 to 0]
  Any Cough | 1 | 0 [0 to 0]
  Severe Cough | 0 | 0 [0 to 0]
  Any Erythema | 0 | 2 [0 to 0]
  Severe Erythema | 0 | 0 [0 to 0]
  Any Pruritis | 3 | 4 [0 to 0]
  Severe Pruritus | 0 | 0 [0 to 0]
  Any Skin Burning Sensation | 1 | 0 [0 to 0]
  Severe Skin Burning Sensation | 0 | 0 [0 to 0]

4. Secondary Outcome: Summary of the Reported Skin/Scalp Irritation Before Treatment and Post-treatment With Either Ivermectin or Placebo (Vehicle Control)
Description: Severe skin/scalp irritations were defined as follows:
  Severe Pruritus - Nearly constant, frequent scratching, very bothersome; Severe Erythema - large areas of the scalp are red; Severe Excoriation - Widespread breaking of the skin involving most of the scalp; Severe Pyoderma - Lesions with crusting or other evidence of infection, involving most of the scalp.
Time Frame: Day 1 up to Day 15 post-application
Population: Skin/scalp irritation was assessed in the Intent-to-treat (Safety) population.
Measure: Number; unit: Participants
Arm/Group | 0.5% Ivermectin | Vehicle Control
Number analyzed (Participants) | 211 | 199
Participants
  Any Pruritus Day 1 (Pre-treatment; N = 211, 199) | 126 | 136 [0 to 0]
  Severe Puritus Day 1 (Pre-treatment; N = 211, 199) | 7 | 10 [0 to 0]
  Any Pruritus Day 2 (N = 210, 199) | 41 | 98 [0 to 0]
  Severe Pruritus Day 2 (N = 210, 199) | 2 | 7 [0 to 0]
  Any Pruritus Day 8 (N = 203, 77) | 31 | 10 [0 to 0]
  Severe Pruritus Day 8 (N = 203, 77) | 0 | 0 [0 to 0]
  Any Pruritus Day 15 (N = 197, 51) | 12 | 3 [0 to 0]
  Severe Pruritus Day 15 (N = 197, 51) | 0 | 0 [0 to 0]
  Any Erythema Day 1 (Pre-treatment; N = 211, 199) | 16 | 23 [0 to 0]
  Severe Erythema Day 1 (Pre-treatment; N= 211, 199) | 0 | 1 [0 to 0]
  Any Erythema Day 2 (N = 210, 199) | 14 | 22 [0 to 0]
  Severe Erythema Day 2 (N = 210, 199) | 0 | 0 [0 to 0]
  Any Erythema Day 8 (N = 203, 77) | 8 | 2 [0 to 0]
  Severe Erythema Day 8 (N = 203, 77) | 0 | 0 [0 to 0]
  Any Erythema Day 15 (N = 197, 51) | 2 | 0 [0 to 0]
  Severe Erythema Day 15 (N = 197, 51) | 0 | 0 [0 to 0]
  Any Excoriation Day 1 (Pre-treatment; N= 211, 199) | 16 | 48 [0 to 0]
  Severe Excoriation Day 1 (Pre-treatment; N=211,199 | 0 | 0 [0 to 0]
  Any Excoriation Day 2 (N = 210, 199) | 14 | 34 [0 to 0]
  Severe Excoriation Day 2 (N = 210, 199) | 0 | 0 [0 to 0]
  Any Excoriation Day 8 (N = 203, 77) | 3 | 8 [0 to 0]
  Severe Excoriation Day 8 (N = 203, 77) | 0 | 0 [0 to 0]
  Any Excoriation Day 15 (N = 197, 51) | 1 | 2 [0 to 0]
  Severe Excoriation Day 15 (N = 197, 51) | 0 | 0 [0 to 0]
  Any Pyoderma Day 1 (Pre-treatment; N = 211, 199) | 0 | 3
  Severe Pyoderma Day 1 (Pre-treatment; N= 211, 199) | 0 | 0
  Any Pyoderma Day 2 (N = 210, 199) | 0 | 3
  Severe Pyoderma Day 2 (N = 210, 199) | 0 | 0
  Any Pyoderma Day 8 (N = 203, 77) | 0 | 1
  Severe Pyoderma Day 8 (N = 203, 77) | 0 | 0
  Any Pyoderma Day 15 (N = 197, 51) | 0 | 0
  Severe Pyoderma Day 15 (N = 197, 51) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the day of application (Day 1) through Day 15 post-application.
Arm/Group | 0.5% Ivermectin | Vehicle Control
Serious Adverse Events (participants affected / at risk) | 0/210 | 0/199
Other Adverse Events (participants affected / at risk) | 0/210 | 0/199

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications